CLINICAL TRIAL: NCT03282864
Title: The Impact of Air Filtration on Health Indicators of Asthmatic Children
Brief Title: The Impact of Air Filtration on Asthmatic Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Underwriters Laboratory, Inc (Unknown); Duke University (Other); Tsinghua University (Other); University of Wisconsin, Madison (Other)
Responsible Party: Principal Investigator, Zhen Li, Attending Physician, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: [2016] 48
Record Dates: First submitted 2017-08-24; First posted 2017-09-14 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Asthma in Children
Keywords: asthma; air pollution; air filtration; indoor air quality; respiratory health
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Every study subject had the air in their bedroom processed by an air filtration device (with a pre-filter, a HEPA filter and an active carbon filter) for two weeks (active comparator arm), processed by a placebo air filtration device (which did not possess the HEPA filter and active carbon filters) for two weeks (placebo arm), and underwent a two-week washout period (no use of air filtration device) between the two intervention periods.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The real air filtration device and the placebo air filtration device looked identical, however the placebo air filtration device lacked the HEPA and active carbon filters which functioned to remove airborne pollutants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bedroom air filtered by an air filtration device (Active Comparator): The air in the bedroom of study subjects in the active comparator arm was filtered by an air filtration device which processed air through a pre-filter, a high efficiency particular air (HEPA) filter and an active carbon filter. The duration of being in the active comparator arm was 2 weeks.
  Interventions: Device: Bedroom air filtered by an air filtration device to remove airborne pollutants
- Bedroom air filtered by a placebo air filtration device (Placebo Comparator): The air in the bedroom of subjects in the placebo arm was filtered by a placebo air filtration device that looked identical to the real air filtration device but did not possess the HEPA filter and the active carbon filter. The duration of being in the placebo arm was 2 weeks.
  Interventions: Device: Bedroom air filtered by an air filtration device to remove airborne pollutants

INTERVENTIONS:
Device: Bedroom air filtered by an air filtration device to remove airborne pollutants — The air in the bedroom of study subjects in the active comparator arm was processed by an air filtration device which pulled air through a pre-filter, a high efficiency particular air (HEPA) filter and an active carbon filter continuously. The air in the bedroom of subjects in the placebo arm was processed by a placebo air filtration device that looked identical to the real air filtration device but did not possess the HEPA filter and the active carbon filter. Each subject was assigned to the active comparator arm and the placebo arm in a randomized order with a two-week washout period scheduled in-between. The subjects, their guardians and the study staff that assessed the health indicators of the subjects were blinded to this order till the end of the study.

SUMMARY:
This study uses a crossover study design to examine the impact of a two-week bedroom based indoor air filtration on the concentration of indoor airborne pollutants, personal exposure to airborne pollutants and health indicators among asthmatic children living in Shanghai, China

DETAILED DESCRIPTION:
This study recruited asthmatic children aged 5 to 14 who were living in Shanghai, China. Every study subject had the air in their bedroom processed by an air filtration device (with a pre-filter, a HEPA filter and an active carbon filter) for two weeks (active comparator arm), processed by a placebo air filtration device (which did not possess the HEPA filter and active carbon filters) for two weeks (placebo arm), and underwent a two-week washout period (no use of air filtration device) between the two intervention periods. The doors and windows of the bedroom were instructed to be kept closed during the intervention periods. The sequence of being in the active comparator arm and the placebo arm was randomized for each subject. The subject, their guardian and researchers who have direct interaction with the study subjects do not know this sequence until after the end of the study.

The study protocol was approved by IRB at Shanghai First People's Hospital, Duke University and University of Wisconsin at Madison. A sample size of 40 was calculated using fractional exhaled nitric oxide (FeNO) as the primary outcome where statistical significance was set at 0.05, power at 90%, and between-subject variance and covariance were estimated from existing literature. Four additional subjects were added to the estimated sample size of 40 to account for potential dropouts. Subjects were recruited from patients who attended the outpatient clinic of the Pediatrics Department of Shanghai First People's Hospital (south section) by Dr. Zhen Li and Dr. Junfeng Zhang's team. Assent was obtained from all study subjects and written informed consent was obtained from their guardians.

During the study, Dr. Michael Bergin's team and Dr. Yinping Zhang's team installed the air filtration devices in the subject's bedroom and measured the indoor concentration, outdoor concentration and personal exposure to airborne pollutants including PM2.5, ozone and volatile organic compounds. Dr. James Schauer's team analyzed the physical, chemical and bioactivity of the airborne particles collected and had no direct contact with the study subjects.

Each subject attended 5 clinical visits at the Shanghai First People's Hospital (South Section) accompanied by their guardian where clinical assessment (of lung function, fractional exhaled nitric oxide, asthma symptom blood draw) was performed by Drs. Zhen Li and Feng Li's team, and the collection of biological media (urine, saliva and nasal fluid) was conducted by Dr. Junfeng (Jim) Zhang's team. In addition, subjects were instructed to measure the peak expiratory flow (PEF) at 7am and 9pm daily and recorded their asthma symptoms at home with the assistance from their guardian(s). The biological media (urine, saliva and nasal fluid) collected was subsequently analyzed by Dr. Junfeng (Jim) Zhang's team for health indicators.

Each subject had access to the result of clinical assessment and health indicator in biological media, as well as free consultation from the medical teams of Drs. Zhen Li and Feng Li. Every subject was remunerated with 1000RMB (equivalent to 152 US dollars) and given a peak expiratory flow meter (worth less than 10 US dollars). All information collected from study subjects were recorded under their subject ID number and kept confidential. Only de-identified data was shared between collaborating investigators. Statistical analysis including mixed-effects models will be conducted on the data collected.

ELIGIBILITY:
Inclusion Criteria:

An eligible child is defined as:

* Aged between 5 and 14
* Have physician-diagnosed asthma
* Had at least one asthma attack during the past year

An eligible household is defined as:

* Has an eligible child
* Located in Shanghai, China

Exclusion Criteria:

* Children who were current smokers or have diseases other than asthma are exclude from study participation

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2017-04-22 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Fractional exhaled nitric oxide (FeNO) | Change of FeNO after the end of the two-week intervention compared to the start of the two-week intervention period
  Fractional exhaled nitric oxide (FeNO) was measured using the NIOX machine

SECONDARY OUTCOMES:
Asthma symptoms | Within 24 hours before the start of intervention and within 24 hours after the end of intervention
  Asthma symptom was evaluated by the Asthma Control Test (ACT) questionnaire
Peak expiratory flow (PEF) | Measured at 7am and 9pm daily during the two-week intervention
  The maximum speed of exhalation (PEF) was measured by a handheld PEF meter (Koka Peak Expiratory Flow Meter)
Lung function | Within 24 hours before the start of intervention and within 24 hours after the end of intervention
  Lung function was assessed by spirometry (Jaeger MasterScreen™ PFT system) and impulse oscillometry (Jaeger MasterScreenTM IOS).

OTHER OUTCOMES:
Malondialdehyde (MDA) concentration in urine | Within 24 hours before the start of intervention and within 24 hours after the end of intervention
  Malondialdehyde (MDA) concentration in urine was measured using the thiobarbituric acid derivatization method and high-performance liquid chromatography (HPLC)
8-OHdG concentration in urine | Within 24 hours before the start of intervention and within 24 hours after the end of intervention
  Concentration of 8-hydroxydeoxyguanosine (8-OHdG) in urine was measured by solid phase extraction and liquid chromatography-mass spectrometry (LC-MS)
Malondialdehyde (MDA) concentration in nasal fluid | Within 24 hours before the start of intervention and within 24 hours after the end of intervention
  Malondialdehyde (MDA) concentration in nasal fluid was measured using the thiobarbituric acid derivatization method and high-performance liquid chromatography (HPLC)
Malondialdehyde (MDA) concentration in saliva | Within 24 hours before the start of intervention and within 24 hours after the end of intervention
  Malondialdehyde (MDA) concentration in saliva was measured using the thiobarbituric acid derivatization method and high-performance liquid chromatography (HPLC)
Interleukin-6 level in saliva | Within 24 hours before the start of intervention and within 24 hours after the end of intervention
  The concentration of interleukin-6 in saliva was measured by enzyme-linked immunosorbent assay (ELISA)
Eosinophil cationic protein concentration in saliva | Within 24 hours before the start of intervention and within 24 hours after the end of intervention
  The concentration of eosinophil cationic protein in saliva was measured by enzyme-linked immunosorbent assay (ELISA)
Blood eosinophil | Only once at the time of enrollment into the study
  Blood eosinophil was assessed using the blood routine test
Allergen profile | Only once at the time of enrollment into the study
  The IgE antibody for 19 allergens were assessed using serum samples from study subjects.
Chemical exposure | During 1 week of the study
  Personal exposure to chemicals including flame retardant and organophosphates was assessed using silicone wristbands that were worn on the wrist of study subjects for 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Michael H. Bergin, PhD, Study Director — Duke University; Junfeng Zhang, PhD, Principal Investigator — Duke University; James J. Schauer, PhD, Principal Investigator — University of Wisconsin, Madison; Yinping Zhang, PhD, Principal Investigator — Tsinghua University; Feng Li, MD, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cui X, Li Z, Teng Y, Barkjohn KK, Norris CL, Fang L, Daniel GN, He L, Lin L, Wang Q, Day DB, Zhou X, Hong J, Gong J, Li F, Mo J, Zhang Y, Schauer JJ, Black MS, Bergin MH, Zhang J. Association Between Bedroom Particulate Matter Filtration and Changes in Airway Pathophysiology in Children With Asthma. JAMA Pediatr. 2020 Jun 1;174(6):533-542. doi: 10.1001/jamapediatrics.2020.0140. PMID 32250418
- [Derived] Brehmer C, Norris C, Barkjohn KK, Bergin MH, Zhang J, Cui X, Teng Y, Zhang Y, Black M, Li Z, Shafer MM, Schauer JJ. The impact of household air cleaners on the oxidative potential of PM2.5 and the role of metals and sources associated with indoor and outdoor exposure. Environ Res. 2020 Feb;181:108919. doi: 10.1016/j.envres.2019.108919. Epub 2019 Nov 13. PMID 31753466